CLINICAL TRIAL: NCT03714880
Title: Cervical Preparation With Mifepristone Prior to Osmotic Dilators: A Randomized, Double-blind, Placebo-controlled Pilot Study
Brief Title: Cervical Preparation With Mifepristone Prior to Osmotic Dilators
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow recruitment compounded by COVID-19
Sponsor: University of California, Davis (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1317056
Record Dates: First submitted 2018-10-17; First posted 2018-10-22 (Actual); Results first posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Second Trimester Abortion
MeSH Terms: interventions — Mifepristone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Mifepristone (Experimental): Participants ingest mifepristone 200 mg oral medication once 18-24 hours prior to dilator placement
  Interventions: Drug: Mifepristone 200 MG
- Placebo (Placebo Comparator): Participants ingest placebo oral medication once 18-24 hours prior to dilator placement
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Mifepristone 200 MG — Ingestion of study medication vs placebo
  Arms: Mifepristone
Drug: Placebo Oral Tablet — Ingestion of study medication vs placebo
  Arms: Placebo

SUMMARY:
The investigators plan to study the role of mifepristone prior to the placement of cervical osmotic dilators to evaluate if the medication helps increase the number of dilators. This may help improve safety of dilation and evacuation (D&E) procedures.

DETAILED DESCRIPTION:
No clear guideline currently exists for best practices involving cervical preparation for women planning dilation and evacuation at 20 weeks and greater. The investigators plan to perform a pilot, randomized, double-blind, placebo-controlled trial. On day 1, 66 participants will receive mifepristone 200 mg orally or placebo 18-24 hours prior to osmotic dilator (Dilapan-S 4-mm) placement (day 2). On day 3, participants will have a D&E procedure. Enrollees will be 18 weeks 0 days to 23 weeks 6 days gestation on the day of the procedure. The primary objective is to evaluate the role of adjunctive mifepristone the day prior to osmotic dilator placement for dilation and evacuation procedures. The primary outcome will be the number of dilators successfully placed. Investigators will compare the number of dilators placed between study arms stratified by gestational age. Secondary outcomes include cervical dilation at time of procedure, proportion of women requiring mechanical dilation at time of surgery, provider impression on ease of procedure and/or difficulty in dilating the cervix when clinically required, and overall complications. Complications or adverse events include cervical laceration requiring repair, perforations, blood transfusions, ED visits, hospitalizations, infection, additional surgical procedures, or extramural deliveries.

ELIGIBILITY:
Inclusion Criteria:

A. Age ≥18 years B. Gestational age to be 18 weeks 0 days through 23 weeks 6 days on procedure date C. Signed informed procedure consent for dilation and evacuation D. Willing to sign informed consent and follow study protocol

Exclusion Criteria:

A. Allergy or known intolerance to mifepristone

B. Known contraindication to mifepristone for cervical preparation prior to dilation and evacuation:

1. Chronic adrenal failure or insufficiency
2. Concurrent use of long-term corticosteroid therapy
3. Inherited porphyrias

C. Any condition that in the opinion of the investigator could impede study participation or collection of study data

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2019-04-26 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Department of Obstetrics and Gynecology, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Mifepristone: Participants ingest mifepristone 200 mg oral medication once 18-24 hours prior to dilator placement
  Mifepristone 200 MG: Ingestion of study medication
- Placebo: Participants ingest placebo oral medication once 18-24 hours prior to dilator placement
  Placebo Oral Tablet: Ingestion of placebo
Period: Overall Study
Arm/Group | Mifepristone | Placebo
Started | 20 | 24
Completed | 19 | 22
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mifepristone | Placebo | Total
Number analyzed (Participants) | 19 | 22 | 41
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 27 [24 to 32] | 27.5 [21 to 30.5] | 27 [24 to 31.5]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Assigned female sex | 19 | 22 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 15 | 17 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 5 | 12
  White | 7 | 11 | 18
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 4 | 2 | 6
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 29.1 [26.4 to 32.6] | 27.9 [23.3 to 32.7] | 28.9 [24.3 to 32.4]
Obstetrical history [Count of Participants; unit: Participants]
  History of vaginal delivery | 11 | 11 | 22
  History of cesarean delivery only | 3 | 4 | 7
  Nulliparous | 5 | 7 | 12
Gestational age [Count of Participants; unit: Participants]
  18w0d-19w6d | 1 | 5 | 6
  20w0d-21w6d | 11 | 9 | 20
  22w0d-23w6d | 7 | 8 | 15
History of cervical procedures [Count of Participants; unit: Participants] | 1 | 1 | 2
Education - high school diploma or less [Count of Participants; unit: Participants] | 9 | 10 | 19
Married, current [Count of Participants; unit: Participants] | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Had Placement of Expected Dilators or More
Description: The number of expected dilators (Dilapan-S) is calculated based on the gestational age. Four dilators are expected to be placed at 18 weeks 0 days to 19 weeks 6 days gestation. Five dilators are expected to be placed at 20 weeks 0 days to 20 weeks 6 days gestation. Six dilators are expected to be placed at 21 weeks 0 days to 21 weeks 6 days gestation. Seven dilators are expected to be placed at 22 weeks 0 days to 23 weeks 5 days gestation. Therefore, at any given gestational age, if the expected number of dilators (or additional dilators) were placed, the participant was counted as "Yes, participant had placement of expected dilators or more."
Time Frame: At time of 1 hour clinic visit (10 minutes)
Measure: Count of Participants; unit: Participants
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 19 | 22
Participants | 17 | 21

2. Secondary Outcome: Cervical Dilation
Description: Measurement of cervical dilation at time of procedure
Time Frame: At time of ~1 hour scheduled procedure time (1 minute)
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 19 | 22
cm | 3.2 [2.6 to 3.6] | 2.6 [2.1 to 3.0]

3. Secondary Outcome: Number of Participants That Required Mechanical Dilation
Description: A count of the number of participants that required of mechanical dilation at time of procedure
Time Frame: At time of ~1 hour scheduled procedure time (10 minute)
Measure: Count of Participants; unit: Participants
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 19 | 22
Participants | 2 | 4

4. Secondary Outcome: Pain Dilator Placement Using Visual Analog Scale
Description: Title: Pain at time of dilator placement. Participants mark their associated pain score on a 10-cm visual analog scale at time of dilator placement with anchors of "no pain" at 0 cm and "worst pain in your life" at 10 cm.
  Higher scores indicate worse outcome.
Time Frame: At time of 1 hour clinic visit (10 minutes)
Measure: Median (Inter-Quartile Range); unit: cm
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 19 | 22
cm | 1.2 [0 to 6.6] | 3.3 [0.6 to 6.1]

5. Secondary Outcome: Provider Assessment of Procedure as "Very Easy" or "Easy"
Description: Survey providers blinded to study grouping regarding overall ease of procedure based on cervical dilation Identified procedures that were categorized as "Very Easy" or "Easy" (Survey response based on Likert scale: "Very Easy," "Easy," "Moderate," "Difficult," "Very Difficult")
Time Frame: At time of ~1 hour scheduled procedure time
Measure: Count of Participants; unit: Participants
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 19 | 22
Participants | 8 | 9

6. Secondary Outcome: Number of Participants That Experienced Complications
Description: Composite of complications including cervical lacerations requiring repair, perforations, blood transfusions, ED visits, hospitalizations, infections, additional surgical procedures, or extramural deliveries
Time Frame: At time of ~1 hour scheduled procedure time (0-30 minute)
Measure: Count of Participants; unit: Participants
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 19 | 22
Participants | 3 | 3

7. Secondary Outcome: Number of Participants That Required Mechanical Dilation
Description: Number of participants that required mechanical dilation at time of procedure
Time Frame: At time of ~1 hour scheduled procedure time
Measure: Count of Participants; unit: Participants
Arm/Group | Mifepristone | Placebo
Number analyzed (Participants) | 19 | 22
Participants | 2 | 4

ADVERSE EVENTS:
Time Frame: 3 days
Arm/Group | Mifepristone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/19 | 1/22
Other Adverse Events (participants affected / at risk) | 0/19 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mifepristone (N=19) | Placebo (N=22)
Elective withdrawal of participant after study medication ingestion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT03714880/Prot_SAP_000.pdf